CLINICAL TRIAL: NCT06916988
Title: Modified Sports Intervention Combined With Context-Focused Intervention in Adolescents With Autism Spectrum Disorder: Protocol for a Mixed Methods Study
Brief Title: Modified and Context-Focused Sports Intervention in Adolescents With Autism: Study Protocol
Acronym: ASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Lidiane Francisca Borges Ferreira, Master in Occupational Studies, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 84826024.6.0000.5149
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Context-centered intervention; Participation; Adolescents; Modified Sports; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Adolescents (n=52) will be randomized into two groups in Phase 1: Sports Stars Brazil (n=26) and Sports Stars Brazil + PREP (n=26). Randomization will occur in blocks, with each randomization taking place once two subgroups of 6-8 participants are recruited.
  A random number generator will be used to create a random sequence of numbers. These numbers will be concealed in individually numbered, opaque, sealed envelopes. This sequence will determine whether participants are assigned to the Sports Stars Brazil group or the control group. A new random sequence will be used for each subgroup randomization until all 52 adolescents are allocated or no additional participants can be recruited.
  Assessors will remain blinded to group allocation. However, due to the nature of the intervention in this study, it will not be possible to ensure blinding for the individuals and intervention therapists.
Who Masked: Outcomes Assessor
Masking Description: Assessors will remain blinded to group allocation. However, due to the nature of the intervention in this study, it will not be possible to ensure blinding for the individuals and intervention therapists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified sports (Placebo Comparator): Control group:
  Modified sports. 26 adolescents performed only the modified sports protocol
  Interventions: Behavioral: Sports Stars Brazil
- Modified sports + context-centered therapy (Experimental): Intervention group:
  Modified sports + context-centered therapy. 26 adolescents performed the modified sports protocol associated with context-centered therapy.
  Interventions: Behavioral: Sports Stars Brazil; Behavioral: context-centered therapy

INTERVENTIONS:
Behavioral: Sports Stars Brazil — Modified sports interventions promote physical activity participation in individuals with ASD by addressing intrinsic factors, however they do not address contextual barriers, such as environmental and interpersonal factors, which also influence participation. Factors like bullying, parents' perceptions often prioritizing therapy intervention, and challenges faced in community programs (as the lack of adaptations in existing programs to meet their needs) are some of these obstacles, which reduce adherence to physical activities (Jachyra et al., 2021). Therefore, it may be necessary to combine interventions targeting intrinsic factors, such as Sports Stars, with those that address the extrinsic contextual factors impacting the participation of adolescents with ASD in their community.
Behavioral: context-centered therapy — The complimentary approach of combining intrinsic (Sports Stars) and extrinsic (PREP) interventions aligns with the relationships between the person, their environment, and the quantity and quality of their participation proposed in the "family of participation related constructs (Imms et al., 2017)." By recognizing that participation depends on both the individual's abilities and the contexts and conditions in which it occurs, professionals can adopt a more holistic and tailored approach to individual needs (Imms et al., 2015).
  Arms: Modified sports + context-centered therapy

SUMMARY:
Adolescents with Autism Spectrum Disorder (ASD) typically engage less in physical activities than their typically developing peers, influenced by intrinsic and extrinsic factors. Modified sports interventions, like Sports Stars Brazil, can improve motor skills and promote lifelong participation in sports by enhancing physical, social, and cognitive abilities. However, adolescents often face barriers to engaging in community sports and recreational activities after completing the program. PREP is an approach designed to address these barriers by modifying environments and empowering families. To date, no study has explored this combination in adolescents with ASD. Objective: This protocol assesses the effectiveness of combining Sports Stars Brazil with PREP to enhance participation and physical literacy in adolescents with ASD and explores participant and family perceptions. Method: A mixed-methods study with two phases: 1) a randomized controlled trial to investigate combined intervention's effects; and 2) evaluation of participant and family perceptions.

DETAILED DESCRIPTION:
Adolescents exhibit higher levels of sedentary behavior compared to other age groups. This situation is even more evident among adolescents with Autism Spectrum Disorder (ASD), who show significantly lower levels of physical activity than typically developing adolescents. Studies have revealed that most adolescents with ASD did not meet the three components of the Canadian 24-Hour Movement Guidelines, which include physical activity, sedentary time, and sleep. Low levels of physical activity may contribute to high rates of physical or mental health problems among young people with ASD, including a higher prevalence of overweight and obesity.

Intrinsic factors, such as mobility limitations and difficulties with social interaction, may restrict the participation of children and adolescents with ASD in physical activities. Despite these challenges, evidence suggests that including these young people in physical activity programs can yield significant benefits, such as increased peer social interaction and improvements in motor and communication skills. However, participation in physical activities tends to decline with age, resulting in less engagement from adolescents with ASD compared to younger children with the same diagnosis. Therefore, it is crucial to develop effective strategies to promote the participation of these individuals in physical activities.

Several interventions aim to promote the participation of children and adolescents with ASD in physical activities, including modified sports programs. These programs are defined as recreational activities where rules, equipment, or spaces are modified to enhance sports inclusion and develop fundamental motor skills. Despite the recognition of the importance of modified sports for children's preparation for sports and physical activity, there is still a lack of such interventions for individuals with disabilities, especially in low- and middle-income countries. To address this gap, the Sports Stars program was developed in Australia. This intervention involves modified sports activities led by professionals and delivered in peer groups. Sports Stars focuses on supporting the development of intrinsic factors, such as physical, social, cognitive, and psychological competence in children, or their physical literacy. The program was adapted to the Brazilian context to promote the participation of children and adolescents with cerebral palsy and ASD in physical activities.

A quasi-experimental study assessed the acceptability and initial outcomes of this modified sports intervention for Brazilian adolescents with ASD. Sports Stars proved to be feasible, and the preliminary results were positive for promoting participation and improving gross motor skills (such as locomotion and object control), physical conditioning, and physical literacy (social, psychological, cognitive, and physical) in these individuals. However, no planned clinical trials have yet been conducted specifically for this population. Although adolescents improved their participation in the Sports Stars program, these individuals and their families still report barriers to participation in sports and community recreational activities.

Modified sports interventions promote participation in physical activities in individuals with ASD by addressing intrinsic factors; however, they do not address contextual barriers, such as environmental and interpersonal factors, which also influence participation. Factors such as bullying, parents' perceptions often prioritizing therapeutic intervention, and challenges faced in community programs (such as the lack of adaptations in existing programs to meet their needs) are still prevalent.

some of these obstacles, which reduce adherence to physical activities. Therefore, it may be necessary to combine interventions targeting intrinsic factors, such as Sports Stars, with those that address the extrinsic contextual factors impacting the participation of adolescents with ASD in their community.

An example of an intervention focused on context is the Pathways and Resources for Engagement and Participation (PREP). PREP is an approach designed for clinicians seeking to increase participation by modifying extrinsic factors or barriers embedded in someone's environment. Examples include physical, social, attitudinal, institutional, and contextual barriers. The main goal is to guide and empower youth and families to solve problems by navigating barriers, sharing the necessary information to help them achieve their desired participation goals. In this approach, the therapist collaborates with the individual and their caregivers to identify facilitators and barriers to participation and create strategies to minimize or remove potential obstacles. A context-based practice study conducted with children with ASD demonstrated that this intervention can promote increased participation in self-chosen activities over time. Furthermore, a feasibility clinical trial showed that the combination of the Sports Stars Brazil and PREP interventions for children with cerebral palsy provided preliminary evidence that this combination led to greater achievement of participation goals and family empowerment compared to Sports Stars alone.

The complementary approach of combining intrinsic interventions (Sports Stars) and extrinsic interventions (PREP) aligns with the relationships between the person, their environment, and the quantity and quality of their participation, as proposed in the "family of constructs related to participation." By recognizing that participation depends on both the individual's skills and the contexts and conditions in which it occurs, professionals can adopt a more holistic and personalized approach to individual needs. Therefore, the objective of this mixed-methods study protocol is to assess the effectiveness of the combined Sports Stars Brazil and PREP intervention for adolescents with ASD in improving participation outcomes (frequency and engagement) and physical literacy (physical, social, cognitive, and psychological competence), as well as to analyze self-perceived performance and satisfaction with the selected physical activity, and the perceptions and experiences of adolescents and their families regarding this combined intervention through qualitative focus groups and photovoice.

Hypotheses:

* Adolescents with ASD who receive the combined Sports Stars Brazil and PREP intervention will demonstrate greater participation in physical activities, and their caregivers will report higher levels of family empowerment, compared to those who receive only Sports Stars Brazil.
* Adolescents who receive the combined Sports Stars Brazil and PREP intervention will exhibit higher levels of physical literacy compared to those who receive only Sports Stars Brazil.

Design This study will be conducted using a mixed-methods approach, combining a randomized clinical trial and two qualitative studies. A central element of the research will be triangulation, which involves applying different analytical techniques to the same data set to assess the validity of the results. This method allows the integration of multiple sources of information, enhancing the comprehensiveness of the findings.

the reliability and robustness of the findings. Consequently, the research incorporates multiple angles of analysis and varied perspectives, ensuring comprehensive results that are not confined to a single approach.

This three-phase study is developed according to the SPIRIT guidelines, which provide guidance for the conduct of clinical trials. Future dissemination of results will be conducted in phase 1 according to the criteria for presenting pilot studies, following the CONSORT guidelines, and in phases 2 and 3 according to the COREQ criteria. The study was approved by the Research Ethics Committee (approval number 84826024.6.0000.5149) and will be registered in Clinical Trials under number XXXX.

Methods Study Design A mixed-methods study consisting of three distinct phases:

* Phase 1: Investigation of the effects of Sports Stars Brazil + PREP compared to Sports Stars alone through a randomized clinical trial (RCT).
* Phase 2: Exploration of caregivers' perceptions regarding their children's experiences using semi-structured focus groups.
* Phase 3: Exploration of adolescents' perceptions and experiences using the photovoice method.

PPI (Public and Patient Involvement) Until the last decade, there were a limited number of studies actively involving individuals with ASD and their families. However, due to the advocacy efforts of patients, families, and activists, as well as the new policy of the journal Autism, which since January 2021 requires authors to report whether individuals with ASD were involved in their work, this number has increased, leading to up to five times more involvement of these individuals in research.

In this approach, public and patient involvement (PPI) occurs "with" or "by" them, rather than being done "for," "about," or "to" them. Researchers, professionals, and the public (patients, caregivers, and representatives of organizations supporting these individuals) will collaborate fully, sharing responsibilities throughout the project, including in the creation of knowledge.

To support this collaboration, the Engagement Matrix (EM) tool will be used. Developed to promote patient involvement in research for those aged 12 and older, the EM is structured with its center focusing on the roles that young people or the public can take on, defined in five distinct roles, and on the practical phases of the project. With the EM as a reference, the principal investigator will be responsible for managing the interactions with the adolescents.Additionally, the tool will enhance collaboration, streamline processes, and allow for more systematic reporting of cooperation.

Two caregivers and two adolescents diagnosed with ASD who have previously participated in Sports Stars Brazil will be invited to join the research team as members. Their participation will be crucial in bringing valuable perspectives and personal experiences that will enrich the development of the project. The most important aspect to consider is that PPI facilitates communication with individuals who have relevant life experiences related to health issues, ensuring that their valuable voices and insights are incorporated/included.

Intervention Phase I: Investigation of the Effects of Sports Stars Brazil + PREP Sports Stars Brazil Group (8 weeks) The intervention will be conducted with groups of 6 to 8 adolescents, lasting 1 hour per day, once a week, for 8 weeks, totaling 8 hours. Each group will be led by a physiotherapist, with the assistance of students and/or professionals in occupational therapy and physical education. Each participant will receive guidance from 1-2 direct and consistent professionals throughout the study. The sessions will be structured in the following order: gross motor skill training (jumping, running, motor control activities using a ball), followed by the introduction of popular sports in Brazil: soccer, handball, basketball, and athletics. Throughout the intervention period, the adolescents will be under the care of pre-trained interventionists. Given that children and adolescents with ASD may exhibit repetitive and stereotypical behaviors, support strategies will be implemented, such as providing verbal feedback, using visual cues, communicating rest times, hydration periods, and activity durations.

Sports Stars + PREP Group (8 weeks) In addition to the Sports Stars program, adolescents randomized to the PREP group will simultaneously receive a context-focused intervention. This intervention aims to identify and remove potential barriers that hinder the participation of adolescents with ASD in sports, as well as recognize facilitators and develop strategies to overcome modifiable barriers. Both interventions will be conducted together by a physiotherapist and a pre-trained occupational therapist. The adolescents will receive personalized support to transition to their preferred physical activity in the community. This support will consist of eight weekly meetings, each approximately one hour long, with a team composed of physiotherapists and occupational therapists.

This intervention will be based on the PREP methodology, which includes five steps: (1) Setting goals, (2) Mapping a plan, (3) Making it happen, (4) Measuring the process and outcomes, and (5) Moving forward.

During this intervention, the therapists, along with the participant and their family/adolescent, will: 1) identify barriers to participating in their preferred physical activities, 2) propose a modification plan, 3) implement modifications to facilitate sports participation, and 4) assess the outcomes of the modifications. This intervention will be conducted individually for each participant, together with their family. The specific type of context-focused intervention and the amount carried out will be recorded by the therapists individually for each participant.

Phase II: Evaluation of Caregivers' Experiences Regarding the Sports Stars Intervention Study Design and Objectives In this phase, a qualitative study will be conducted with the aim of exploring the experiences of family members of adolescents with ASD who participated in the Sports Stars program.

Procedures and Data Collection

Data collection for Phase II will occur as follows:

After participation in the Sports Stars Brazil + PREP intervention, focus groups will be held with one family member of each participant at the School of Physical Education, Physiotherapy, and Occupational Therapy of UFMG. Data will be collected in each focus group only once and in person, with an expected duration of 1 hour per interview, extendable if necessary. To ensure homogeneity in data collection, the interviewers responsible will undergo prior training.

Sample characterization data, which are considered important for this study, will be collected before the focus groups and will include: age, gender, communication level classification (for adolescents), socioeconomic status, and parents' education level. During the interview, only the adolescents and interviewers will be present. Semi-structured questions will be asked, focusing on the Family Participation Constructs, which provide the theoretical framework for the Sports Stars and PREP interventions. Additionally, parents will be asked about their experiences participating in the combined Sports Stars Brazil and PREP program.

During the focus groups, the interviewers will present an explanatory video on the "Family of Participation Constructs" (https://www.youtube.com/watch?v=NLzQW2R9XAM), produced by the researchers. This video will highlight the key aspects of the Participation domain of the International Classification of Functioning, Disability, and Health (ICF) in a familiar language, to help clarify the discussion on experiences in the combined Sports Stars Brazil + PREP program.

The focus groups with parents will be conducted immediately after the intervention and will be recorded for later transcription and data analysis. The audio of the focus groups will be recorded for later transcription. After this process, the interviewee will have access to the transcription to verify the data and information before content analysis by the researchers. Additionally, during the focus groups and facilitation, if deemed necessary by the evaluator, notes will be taken. For qualitative data analysis, the MAXQDA software will be used.

Phase III: Evaluation of Adolescents' Experiences Regarding the Sports Stars Intervention Through Photovoice Study Design and Objectives In this phase, a qualitative study will be conducted using the Photovoice method, with the aim of exploring the experiences of adolescents with ASD who participated in the Sports Stars program. Photovoice is a useful tool for adopting a participant-centered strategy, focusing on participation and individual perceptions.

Procedures and Data Collection

Data collection for Phase III will occur as follows:

The third initial phase of the study will be structured in six distinct stages and will begin in the fourth week of the intervention.

Photography Training: Adolescents, accompanied by a responsible adult, will receive basic training in photographic techniques and camera (or smartphone) use. This training will also address ethics and consent. To ensure homogeneity in data collection, the interviewers will undergo prior training.

Image Collection: The adolescents will be instructed, through guided questions, to capture 18 photos representing their participation, with 3 photos for each question.

The activity will take place over 45 days, allowing the adolescents to reflect on their involvement in various aspects of daily life.

Reflection on the Images: After the photo collection, the adolescents will meet with a trained evaluator for an interview to reflect on their images. Each photo will be discussed, and the adolescents will describe their narratives or captions, explaining the meaning behind their choices.

Transcription and Categorization: The focus groups will be transcribed and categorized to facilitate data analysis.

Validation of Results: The results will be discussed and validated with caregivers.

Presentation of Results: The findings will be presented to professionals, families, and the community, promoting the exchange of experiences and learnings.

This process aims not only to document the adolescents' experiences but also to encourage deep reflection on their lives and foster enriching dialogue. A study demonstrated that Photovoice is highly valued by adolescents aged 15 to 17 who use mental health services. This approach promotes personal reflection, the identification of strengths, and the increase of empowerment, which is the main goal of Photovoice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD).
* Level I of functioning (able to maintain interaction and adapt to changes).
* Level II of functioning (able to communicate with others but faces difficulties when changes occur) according to the Autism Spectrum Disorder Social Communication Functioning Classification System.

Exclusion Criteria:

* Cognitive limitations
* Behavioral limitations
* Clinical limitations (e.g., severe cardiorespiratory disease)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Physical Literacy Profile Questionnaire | From registration to end of treatment in 10 weeks
  As an outcome measure, the Physical Literacy Profile Questionnaire will be used, currently being validated by our research group. Developed in Portuguese, this instrument assesses the level of Physical Literacy in children, adolescents, and adults (ages 6-21), focusing on the individual's perception of their participation in the Sports Stars (SS) program. The questionnaire consists of two parts: the first, with 5 questions, evaluates the participant's perception of their experience in the modified sports program; the second, composed of 24 multiple-choice items, examines the individual's performance in physical, social, and cognitive skills. Each item is rated on a scale of 0 to 2 (0: does not perform, 1: performs partially, 2: fully performs). Higher scores (closer to 2) indicate better physical literacy and greater engagement, while lower scores (closer to 0) suggest poorer outcomes.
Goal Attainment Scale | From registration to end of treatment in 10 weeks
  Goal Attainment Scale : A scale used to assess and quantify the achievement of goals previously established in collaboration with the patient/family. This allows for the evaluation of goal attainment and comparison of the interventions used in the process. The scores range from (+2) for the best outcomes to (-2) for the worst, in accordance with the expected results. It is recommended to set at least two goals and a maximum of four to be achieved within the same period. Higher scores (closer to +2) represent better outcomes, indicating that the goal was successfully achieved or even exceeded. Conversely, lower scores (closer to -2) indicate worse outcomes, suggesting that the goal was not achieved as planned.
Canadian Occupational Performance Measure | From registration to end of treatment in 10 weeks
  Canadian Occupational Performance Measure: A widely used assessment tool designed to measure a person's perceived performance and satisfaction with their daily activities (occupations). It allows individuals to identify and prioritize the areas in which they want to see improvement.
  The COPM uses a 10-point scale for both performance and satisfaction, with scores ranging from 1 to 10. A score of 1 indicates "not able to perform" or "extremely dissatisfied," while a score of 10 indicates "able to perform at the desired level" or "extremely satisfied." Higher scores indicate better outcomes, meaning greater satisfaction and higher perceived performance in the selected activities.
Family Empowerment Scale | From registration to end of treatment in 10 weeks
  The Family Empowerment Scale is an assessment tool used to measure the empowerment of families with children who have disabilities. It evaluates how well families feel they can influence decisions regarding their child's care and the services they receive. The scale focuses on key areas such as family support, decision-making, and advocacy.
  The FES uses a 5-point Likert scale, with scores ranging from 1 to 5. A score of 1 indicates strong disagreement or low empowerment, while a score of 5 indicates strong agreement or high empowerment. Higher scores represent better outcomes, indicating greater family empowerment, with families feeling more confident and capable in managing their child's needs and advocating for services.

CONTACTS AND LOCATIONS:
Overall Officials: Hércules R Leite, Doctor, Study Director — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
Sharing of individual participant data will not be carried out due to privacy and confidentiality concerns.

REFERENCES:
- [Background] Fernandes AC, Souto DO, de Sousa Junior RR, Clutterbuck GL, Wright FV, de Souza MG, Ferreira LFB, Cardoso Rodrigues AA, Camargos ACR, Leite HR. Sports Stars Brazil in children with autism spectrum disorder: A feasibility randomized controlled trial protocol. PLoS One. 2023 Nov 8;18(11):e0291488. doi: 10.1371/journal.pone.0291488. eCollection 2023. PMID 37939077